Household Income and Child Development in the First Years of Life (Baby's First Years) NCT 03593356

Consent Form for current wave of age-6 assessments IRB Approval Date: June 14, 2024



Research Consent Form (Page 1)

Attached to Protocol: TC IRB 18-210
IRB Protocol Title: Baby's First Years

Principal Investigator: Kimberly Noble, MD, PhD

Participation Duration: Six Years
Anticipated Number of Participants: 1,000

Study Sponsor(s): National Institute of Child Health and Human Development, private foundations

| Contact | Title | Contact Type | Number |
|----------------|------------------|------------------------|----------------|
| Kimberly Noble | MD, PhD | Principal Investigator | (212) 678-3486 |
| Lauren Meyer | Project Director | Administrative | (608) 291-7359 |

### Key Information about this research

The goal of this research study is to gain an understanding of the role of family experiences on young children's development. Both your and your child's participation in this study is voluntary. There are no direct benefits from participating in this research study, although this study may be helpful in understanding the factors that affect how children learn and grow. The risks for participating are minimal: the primary risks are unlikely disclosure of personal information and possible mild irritation from the EEG cap. If at any time you or your child wish to take a break, you are free to do so.

This study is sponsored by National Institute of Child Health and Human Development and national and local private foundations.

### Invitation to participate in the Baby's First Years 6th Year Visit

You have agreed to participate in the research study called Baby's First Years. We want to understand the role of experience on young children's development. Your decision to participate in the 6<sup>th</sup> year visit will <u>not affect</u> the 4MyBaby card monthly gift you are receiving from the study. You will continue to receive the monthly gift until 3 months after your child's sixth birthday even if you decide not to participate in this interview.

The things we will ask you to do during this 2.5 - 3-hour visit

# You will have the opportunity to...

- Take a survey: answer questions about you, your family, household income/finances; how you have been feeling lately; and the last year of your child's life
- Complete iPad activities: short games to measure attention and sorting

### Your child will have the opportunity to...

- Play a few iPad games and other games: these activities will measure your child's developing skills. In order to use one of the games we will be playing with you and your child, non-personally identifiable information such as birth month and year, race, ethnicity, education level, and gender will be shared with the operator of the app
- **Have an EEG measurement:** during this measurement, your child will wear a child-friendly cap with sensors that can view and record brain activity
- **Donate nails:** we will invite your child to provide a nail sample (collected by cutting) to measure stress levels in the body

Both you and your child will have the opportunity to...

Teachers College, Columbia University Institutional Review Board

Protocol Number: 18-210

Consent Form Approved Until: 09/07/2024



- Play together: we will observe and videotape you and your child participating in some activities
- **Donate saliva:** by swabbing the inside of the cheek and gums with a cotton swab, to help us better understand how life experiences show themselves in the body
- Measure your height and weight

You can skip any parts of the visit in which you do not want to participate or skip any questions that you do not want to answer.

### **Voluntary Participation**

Participating in this study is voluntary. Even if you decide to be part of the study now, you may change your mind and stop at any time. You do not have to answer any questions you do not want to answer. If you decide to withdraw before this study is complete, your data will be kept confidential. You can participate in the research even if you do not want your child to participate, and you can indicate that you would like your child to participate even if you do not want us to collect any information from you.

If at any time you or your child would like to stop or take a break (e.g. a break for eating or rest) you are free to do so.

We may contact you for future waves of data collection. You have the right to decline to participate at any time.

#### **Risks and Burdens**

Risks of participating in this research study to you or your child are minimal.

**General risks:** Although rare, one risk of participation in this study is from accidental disclosure of your research information. To address this potential risk, all written identifying information about you is stored in a locked desk drawer. Any electronic or digital information will be stored on a computer that is password protected. All data are encrypted and stored securely to help protect your privacy.

Additionally, you may find some of the questions asked to be too personal, embarrassing or sensitive. You may skip any questions that you do not wish to answer.

**EEG and saliva and nails donation risks:** The risks associated with using the EEG device with children are minimal and may include some discomfort and mild skin irritation or redness. Risks involved with saliva collection may include mild discomfort. We use certified medical grade equipment which has been safely utilized with children. Risks involved with nails collection may include mild discomfort. We use equipment safely utilized with children and thoroughly sanitized following each use.

**Audio/Video recording risks:** If you consent to be audio/video recorded or photographed in today's research session there is a potential risk of a loss of confidentiality in your research participation. The research team maintains strict data privacy standards to ensure your personal details and responses are de-identified. Additionally, you may withdraw permission to audio/video record or photograph at any time.

You are free to stop, skip, or take a break from any part of the research session at any time.

**Benefits:** There are no direct benefits from participating in this research study. This study may be helpful in understanding the factors that affect how children learn and grow.

## Confidentiality

Researchers will keep all of your personal data private and secure. Only the study team and members of the Teachers College

Teachers College, Columbia University Institutional Review Board

Protocol Number: 18-210

Consent Form Approved Until: 09/07/2024



Institutional Review Board (IRB) may review identifiable data that you provide as part of this study. Otherwise, all information obtained from your participation in this study will be held strictly confidential and will be disclosed only with your permission or as required by U.S. or State law.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers with this Certificate may not disclose or use information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information protected by this Certificate **cannot** be disclosed to anyone else who is not connected with the research **except**:

- if you have consented to the disclosure;
- if it is used for other scientific research, as allowed by federal regulations protecting research subjects; or
- if there is a federal, state, or local law that requires disclosure. For example:
  - o your personal information may be disclosed if we learn that you or someone else is at high or imminent risk of harm.
  - your personal information may be disclosed if we learn of possible abuse of a minor. If a child is in danger of abuse, neglect, or endangerment, we are obligated to report this information to child protection authorities. If this happens, we will take steps to ensure safety of those indicated.

The researchers plan to publish the results of this study. To protect your privacy, they will not include any information that could directly identify you. Your name will never appear in any publication. Your deidentified information collected in this study may be used for future research studies and will be shared, without your name or any other identifying data attached, with a bank of data maintained at the University of Michigan. This bank is called the Inter-University Consortium for Political and Social Research (ICPSR). The data in this bank can be used by researchers at other institutions besides this one, but the data you have provided can never be traced back to you.

A description of this study will be posted on a public website, http://ClinicalTrials.gov, and summary results of this study will be posted on this website at the conclusion of the research, as required by the National Institutes of Health (NIH), the study sponsor. No information that can identify you will be posted.

After completing the visit, the information that you provide will be transferred to a secure storage platform at Teachers College, Columbia University and the University of Wisconsin. The files linking your name to the participant number will be kept in a password-protected database to which only key research staff will have access.

**Saliva and nails:** Saliva and nail samples will be mailed without any identifying information to a lab for chemical analysis, and then destroyed. Biospecimens, like saliva, that are collected as part of this study **will not** be used for commercial profit, and analysis **will not** include whole genome sequencing. Biospecimens will be destroyed once they are processed for this study, and **will not** be used in future research studies.

## **Video Recording**

The purpose of the video- and audio-recorded playtime activity is to understand the different ways in which mothers interact with their children and the kinds of language that children are using. The digital audio and video files are stored on a password protected computer, and will be handled in the same way as the other identifiable information collected in this study (see the "Confidentiality" section for more information). No information that can identify you will be posted publicly. The audio and video files will be stored indefinitely, but you can request for them to be deleted at any time.

In addition to the playtime activity, we may request for parts of the visit to be recorded for quality control purposes only. If you do not wish to be recorded, you may opt out.

Teachers College, Columbia University Institutional Review Board

Protocol Number: 18-210

Consent Form Approved Until: 09/07/2024



| Compensation |
|---|
| For your participation in the research session today you will receive payment and a small toy as a gift for your child. Your compensation is not contingent on completing the study. \$\Begin{align*} \pmu \text{200}: For the in-person visit \end{align*} |
| □ +\$10: For keeping the originally scheduled appointment |
| In some limited circumstances, the visit will be split and the survey will be offered via phone in advance of the university visit: \$\Begin{align*} \$100: For the survey (when completed via phone) \\ \$150: For the in-person visit (when following a phone survey) \\ \$\Begin{align*} +\$10: For keeping the originally scheduled in-person appointment |
| Transportation |
| The study team will arrange round-trip car services for your transportation to the university office for your visit. |
| If you decline car service, you will be paid if you travel on your own. Payment for travel is dependent upon mileage distance (round trip) from your home to the study site as follows: \$30 for 1-40 miles round trip, \$55 for 41-80 miles round trip, \$80 for 81-120 miles round trip, \$110 for 121-160 miles round trip. If your start and end points are different, that is okay; we pay for the total miles driven. We will help you calculating the estimated drive. The rates are at or above the current IRS mileage reimbursement rate of 67 cents per mile. If you live farther than 80 miles away, we will make individual arrangements with you. |
| Who to Contact |
| If you have any questions or concerns about the study, you may contact principal investigator: Kimberly Noble, kgn2106@tc.columbia.edu, (212) 678-3486 or the project director: Lauren Meyer, bfystudy@gmail.com, (608) 291-7359. |
| If you have questions or concerns about your rights as a participant: There is a group of people, called an Institutional Review Board, organized to protect the rights and welfare of people involved in research. |
| Contact the Teachers College Institutional Review Board at: 525 W 120th St, New York, NY 10027 Telephone: (212) 678-3000 Email: irb@tc.edu |
| Statement of Consent |
| I have reviewed the consent form including the purpose, procedures, risks, benefits, and alternatives with the researcher. Any questions I had were answered to my satisfaction. I am aware that by agreeing to continue, I am agreeing to take part in this research study and to be contacted for future study opportunities. I am not waiving (giving up) any of my legal rights by signing this consent form. I will be given a copy of this consent form to keep for my records. |
| Signature |
| Parent/Guardian Print NameDate |

Teachers College, Columbia University Institutional Review Board

Protocol Number: 18-210 Consent Form Approved Until: 09/07/2024





| Researcher | | |
|------------|------------|------|
| Print Name | _Signature | Date |

Teachers College, Columbia University Institutional Review Board

Protocol Number: 18-210 Consent Form Approved Until: 09/07/2024